CLINICAL TRIAL: NCT01158092
Title: A Randomized Controlled Trial Comparing Cooled Radiofrequency Denervation to Conservative Treatment as a Treatment for Sacroiliac Joint Pain Using the SInergy™ System
Brief Title: Trial Comparing Treatment With SInergy™ System to Conservative Treatment for Chronic Sacroiliac Joint Pain
Acronym: SI-RCT-Ross
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Baylis Medical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BMC-SI-CIP-002
Record Dates: First submitted 2010-07-06; First posted 2010-07-08 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Chronic Sacroiliac Joint Pain
MeSH Terms: interventions — Therapeutics; Conservative Treatment

ARMS (2):
- Treatment with SInergy™ System (Active Comparator): Lateral branch denervation using the SInergy™ System
  Interventions: Device: Treatment with SInergy™ System
- Conservative Treatment (Active Comparator): Treatment with physical therapy, chiropractic care, and medication
  Interventions: Other: Conservative Treatment

INTERVENTIONS:
Device: Treatment with SInergy™ System — Lateral branch denervation using the SInergy™ System
  Arms: Treatment with SInergy™ System
Other: Conservative Treatment — Treatment with physical therapy, chiropractic care, and medication
  Arms: Conservative Treatment

SUMMARY:
The purpose of this study is to evaluate the effectiveness of cooled radiofrequency denervation of the sacroiliac region using the SInergy System compared to conservative treatment in the treatment of sacroiliac joint pain.

ELIGIBILITY:
Inclusion Criteria:

* Predominantly axial pain below the L5 vertebrae
* >75% pain relief from 2 separate lateral branch blocks done on different days (followed by return to baseline pain)
* Chronic axial pain lasting for longer than six months: 3 day average VAS between 4 and 8.
* Age greater than 18 years.
* Failed to achieve adequate improvement with comprehensive non-operative treatments, including but not limited to: activity alteration, non-steroidal anti-inflammatory, physical and/or manual therapy, and fluoroscopically guided steroid injections in and around the area of pathology.
* All other possible sources of low back pain have been ruled out, including but not limited to: the intervertebral discs, bone fracture, the zygapophyseal joints, the hip joint, symptomatic spondylolisthesis, tumor and other regional soft tissue structures (this is done by physical exam, medical history, and MRI/CT/X-ray as required)

Exclusion Criteria:

* Beck Depression Score >20 or irreversible psychological barriers to recovery
* Spinal pathology that may impede recovery such as spina bifida occulta, spondylolisthesis at L5/S1, or scoliosis.
* Moderate or severe foraminal or central canal stenosis
* Systemic infection or localized infection at anticipated introducer entry site.
* Concomitant cervical or thoracic pain greater than 2/10 on a VAS
* Uncontrolled or acute illness
* Chronic severe conditions such as rheumatoid/inflammatory arthritis
* Pregnancy
* Active radicular pain
* Immunosuppression (eg. AIDS, cancer, diabetes, surgery <3 months ago)
* Worker's compensation, injury litigation, or disability remuneration
* Allergy to injectants or medications used in procedure
* High narcotics use (>30 mg hydrocodone or equivalent)
* Patients who smoke. Termination for at least 6 months and no smoking during follow up period are acceptable with caution.
* Body Mass Index greater than 29.9 (obese).
* Subject unwilling to consent to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2010-07; Primary Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Pain status change for sacroiliac region pain intensity assessed using visual analogue scale (VAS) | 12 months

SECONDARY OUTCOMES:
Change in bodily pain evaluated using SF-36 Bodily Pain | 12 months
Change in physical functioning evaluated using SF-36 Physical Function | 12 months
Change in disability evaluated using Oswestry Disability Index 2.0 | 12 months
Change in quality of life using the Assessment of Quality of Life (AQOL) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Edgar L Ross, M.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital Pain Trials Center, Chestnut Hill, Massachusetts, United States